CLINICAL TRIAL: NCT01195441
Title: Prediction and Prevention of Preeclampsia by First Trimester Ultrasound
Acronym: Screen-tox
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EUDRACTNUMMER 2009-017833-23; 2009-017833-23 (EudraCT Number)
Record Dates: First submitted 2010-09-01; First posted 2010-09-06 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Doppler ultrasound; First trimester; Acetylsalicylic acid
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether the Fetal Medicine Foundation algorithm for individual risk calculation for preeclampsia (PE) and pregnancy induced hypertension (PIH) is suitable to identify women in high risk of developing these diseases in a Norwegian population.

DETAILED DESCRIPTION:
It has been shown that low dose acetylsalicylic acid (ASA) in pregnancy reduces adverse outcome of pregnancy in women that have high risk of developing preeclampsia (PE). It is a challenge for the clinician to identify the high risk women. Doppler blood flow measurements in uterine arteries in second trimester have been shown useful to predict the development of the disease but prophylactic treatment with ASA from this point in pregnancy has not been proven effective. Fetal Medical Foundation has developed an algorithm that calculates individual risks for PE/ PIH based on Doppler blood flow measurements and anamnestic information.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Nulliparous
* Para 1+ with previous preeclampsia or gestational hypertension
* last menstrual period (LMP) pregnancy length at inclusion < 13 weeks
* Residence in Trondheim + 8 surrounding municipalities

Exclusion Criteria:

* Pregnancy length > 13+6 weeks (CRL > 85 mm)
* Twins
* Missed abortion
* Fetal anomaly

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Development of preeclampsia | september 2012
Onset time of preeclampsia | September 2012

SECONDARY OUTCOMES:
Gestational age at delivery | September 2012
Number of induction of deliveries due to preeclampsia | September 2010
Number of instrumental deliveries due to preeclampsia | September 2012
Perinatal morbidity | September 2012
Maternal morbidity | September 2012

CONTACTS AND LOCATIONS:
Overall Officials: Ragnhild B Skraastad, Cand Med, Principal Investigator — LBK, NTNU, National Center for Fetal Medicine; Kjell Aa Salvesen, Dr Med, Study Director — LBK, NTNU, National Center for Fetal Medicine; Harm-Gerd K Blaas, Dr Med, Study Director — LBK, NTNU, National Center for Fetal Medicine
Locations (1):
- National Center for Fetal Medicine, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Skrastad RB, Hov GG, Blaas HG, Romundstad PR, Salvesen KA. Risk assessment for preeclampsia in nulliparous women at 11-13 weeks gestational age: prospective evaluation of two algorithms. BJOG. 2015 Dec;122(13):1781-8. doi: 10.1111/1471-0528.13194. Epub 2014 Dec 4. PMID 25471057
- [Result] Skrastad RB, Hov GG, Blaas HG, Romundstad PR, Salvesen KA. A prospective study of screening for hypertensive disorders of pregnancy at 11-13 weeks in a Scandinavian population. Acta Obstet Gynecol Scand. 2014 Dec;93(12):1238-47. doi: 10.1111/aogs.12479. Epub 2014 Sep 17. PMID 25146367